CLINICAL TRIAL: NCT05855161
Title: Effectiveness of Rebound Therapy on Balance and Gait in Parkinson's Patients
Brief Title: Effectiveness of Rebound Therapy in Parkinson's Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sefa Eldemir, Principal Investigator, Cumhuriyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5-PD-Rebound therapy-RCT
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; rebound therapy; task oriented training; balance and walking performance
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Two groups as rebound group and control group
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rebound therapy (Experimental): The group that will perform exercises on a trampoline.
  Interventions: Other: Rebound therapy
- Control group (Experimental): The group that will perform exercises on a stable surface.
  Interventions: Other: Exercises on a stable surface

INTERVENTIONS:
Other: Rebound therapy — Participants will receive exercise-based training on a trampoline
  Arms: Rebound therapy
Other: Exercises on a stable surface — Participants will receive exercise-based training on a stable surface
  Arms: Control group

SUMMARY:
Today, physiotherapy approaches in Parkinson's Disease (PD) form the basis of optimal treatment together with medical and surgical treatment. It is stated that various rehabilitation interventions may be effective in the field of physiotherapy. The frequently preferred among these rehabilitation interventions is the conventional treatment approach. In the conventional treatment, various exercises are preferred to improve balance and walking, as well as stretching and strengthening. On the other hand, rebound therapy require strong integration of the neuromuscular system and provide more active use of lower extremity muscle strength. Rebound therapy have been shown to be effective in improving balance in many neurological disease groups, but there is very little study on rebound therapy in PD. It was shown that rebound therapy improve proprioceptive sense, joint range of motion and quality of life. On the other hand, no study has been found showing its effect on balance and walking. Therefore, there is a need to investigate the effectiveness of rebound therapy on balance and walking.

DETAILED DESCRIPTION:
This study is a randomized controlled study. The patients will be randomly divided into two groups as rebound and control. The rebound group will perform exercises on a trampoline, consisting of 15 minutes of trunk and extremity stretching, 10 minutes of walking, and approximately 30 minutes of task-oriented exercises, twice a week for six weeks. While the control group will follow the same program as the rebound group, they will only perform task-oriented exercises on a stable surface, unlike the rebound group. As the outcome measures, disease severity and disability, balance, and gait performance will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 40-80 years of age
* Having diagnosed with "Parkinson's Disease" by a specialist physician
* Having between 1-3 stages according to the Hoehn and Yahr Scale
* Mini-Mental Test score more than or equal 24

Exclusion Criteria:

- Any orthopedic, vision, hearing, cardiovascular, or perception problems that may affect the research results

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Static Balance- Baseline | Assessment will be conducted before the intervention
  Assessment will be made with the Biodex Balance System
Static Balance- Post intervention | Assessment will be conducted immediately after the intervention
  Assessment will be made with the Biodex Balance System
Gait speed- Baseline | Assessment will be conducted before the intervention
  Assessment will be made with the BTS G-Walk, (BTS SpA, Via della Croce Rossa, 11 Padova, Italy; SN: 0213-0378) during gait
Gait speed- Post intervention | Assessment will be conducted immediately after the intervention
  Assessment will be made with the BTS G-Walk, (BTS SpA, Via della Croce Rossa, 11 Padova, Italy; SN: 0213-0378) during gait
Knee strength- Baseline | Assessment will be conducted before the intervention
  Assessment will be made with an isokinetic dynamometer (Cybex Humac Norm Testing and Rehabilitation System, CSMI, USA)
Knee strength-Post intervention | Assessment will be conducted immediately after the intervention
  Assessment will be made with an isokinetic dynamometer (Cybex Humac Norm Testing and Rehabilitation System, CSMI, USA)

CONTACTS AND LOCATIONS:
Locations (1):
- Sivas Cumhuriyet University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Sivas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to make PD data but when the statistical analysis of all data is made, all results will be shared.

REFERENCES:
- [Background] Daneshvar P, Ghasemi G, Zolaktaf V, Karimi MT. Comparison of the Effect of 8-Week Rebound Therapy-Based Exercise Program and Weight-Supported Exercises on the Range of Motion, Proprioception, and the Quality of Life in Patients with Parkinson's Disease. Int J Prev Med. 2019 Aug 12;10:131. doi: 10.4103/ijpvm.IJPVM_527_18. eCollection 2019. PMID 31516672
- [Derived] Eldemir S, Polat EA, Gokdogan CM, Eldemir K, Guclu-Gunduz A, Yilmaz R, Akbostanci MC, Yazici G. The effect of rebound therapy in Parkinson's disease: A single-blinded randomized controlled trial. Gait Posture. 2026 Jan 25;125:110105. doi: 10.1016/j.gaitpost.2026.110105. Online ahead of print. PMID 41592453